CLINICAL TRIAL: NCT07035509
Title: Randomized Control Study on Normal Saline vs Plasmalite vs Plasma in REsuscitation of SEpsis Trial (RESET) - A Feasibility and Comparative Study
Brief Title: Randomized Control Study in REsuscitation of SEpsis Trial
Acronym: RESET
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Fundación Cardioinfantil Instituto de Cardiología (Other)
Collaborators: University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEIC-456-2024
Record Dates: First submitted 2025-03-04; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Septic Shock; Pediatric Critical Illness
Keywords: sepsis; Septic shock; Fluid bolus; plasma; pediatric; crystalloids
MeSH Terms: conditions — Shock, Septic; Sepsis | interventions — Saline Solution; Ringer's Lactate

STUDY DESIGN:
Intervention Model Description: Patients diagnosed with septic shock who meet the inclusion criteria will be randomly assigned to one of three intervention arms:
  * Group 1: Bolus dose of 10 mL/kg normal saline (NS) (max. 500 mL) administered over <15 minutes.
  * Group 2: Bolus dose of 10 mL/kg Ringer's lactate (max. 500 mL) administered over <15 minutes.
  * Group 3: Pharmaceutical fresh frozen plasma (OCTAPLAS LG®), bolus dose of 10 mL/kg (max. 500 mL) administered over <15 minutes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- OCTAPLAS LG (Experimental): Pharmaceutical fresh frozen plasma (OCTAPLAS LG®), bolus dose of 10 mL/kg (max. 500 mL) administered over <15 minutes
  Interventions: Biological: Pharmaceutical fresh frozen plasma
- Normal saline (Active Comparator): Bolus dose of 10 mL/kg normal saline (NS) (max. 500 mL) administered over <15 minutes.
  Interventions: Drug: Normal Saline
- Ringer Lactate (Active Comparator): Bolus dose of 10 mL/kg Ringer's lactate (max. 500 mL) administered over <15 minutes.
  Interventions: Drug: Ringer lactate (RL)

INTERVENTIONS:
Biological: Pharmaceutical fresh frozen plasma — OCTAPLAS LG® has been registered with INVIMA in Colombia for five years and is used as a plasma replacement in cardiac surgery, hematologic diseases, or intensive care settings where blood bank plasma is unavailable
  Arms: OCTAPLAS LG
Drug: Normal Saline — Bolus dose of 10 mL/kg normal saline (NS) (max. 500 mL) administered over <15 minutes.
  Arms: Normal saline
Drug: Ringer lactate (RL) — Bolus dose of 10 mL/kg Ringer's lactate (max. 500 mL) administered over <15 minutes.
  Arms: Ringer Lactate

SUMMARY:
Crystalloids vs. Synthetic Plasma for Fluid Resuscitation in Children with Sepsis - REsuscitation of SEpsis Trial (RESET): A Comparative and Feasibility Study This research study, called the REsuscitation of SEpsis Trial (RESET), is a randomized clinical trial comparing crystalloids and synthetic plasma for fluid resuscitation in children with sepsis. Below, we explain some key aspects you should be aware of.

What is a Clinical Trial? A clinical trial is a type of medical research designed to gather more information on how our bodies respond to medications or other treatments.

Most new medical treatments must be evaluated in clinical trials before they can be approved by government agencies. These agencies ensure that new treatments are not only safe but also beneficial for patients-what medicine refers to as being "safe and effective." If a new treatment has not yet been approved, it is considered "experimental."

Researchers analyze the results of multiple clinical trials to determine which medications work best and how they function. The advancement of medical science requires the participation of many people in numerous studies worldwide.

What is the Purpose of This Study? This study evaluates whether Octaplas LG helps children and adolescents with sepsis and whether it improves the function of blood vessels inflamed due to infection. Sepsis occurs when an infection severely affects a person's health.

Octaplas LG is a medication approved for use in Colombia. It is known as pharmaceutical plasma and is obtained from voluntary donors worldwide. It undergoes an ultra-detailed sterilization process using the most advanced techniques for processing blood derivatives. In medicine, fresh frozen plasma (FFP) is typically used, which is the equivalent of Octaplas LG but with far fewer industrial sterilization processes. These additional processes in Octaplas LG significantly reduce the risk of transmitting infections.

Although Octaplas LG is approved by INVIMA, its use for fluid resuscitation has not yet been approved.

This study will compare Octaplas LG with normal saline solution and Ringer's lactate, which are commonly used for rehydrating patients. All three treatments will be administered in the same manner.

Why is My Child Being Asked to Participate?

Your child is being invited to participate in this clinical study because:

They are receiving care in the pediatric intensive care unit (PICU). They are between one month and 18 years old. They have been diagnosed with sepsis and require fluid resuscitation. Your child's participation is voluntary. If you decide not to participate, your child will not lose any medical benefits. Your child's doctor has determined that they may be a good candidate for this study. You are free to discuss participation with your family, friends, or another physician.

Some members of your child's healthcare team may also be involved in this research. They are dedicated to your child's care as well as the objectives of this study. However, you are not obligated to participate. If you choose to enroll your child, you will be asked to sign an informed consent form.

How Will My Child Be Assigned to a Treatment Group? Upon admission to the pediatric intensive care unit (PICU), if your child has a confirmed sepsis diagnosis and requires intravenous fluids or plasma to support heart function, they will be randomly assigned to one of the three treatment groups.

Randomization is a research method used in clinical trials to assign patients to study groups in an unbiased way-similar to drawing numbers from a hat. Neither you, your child's doctor, nor the researchers will choose which group your child is placed in. Instead, a computer will randomly assign them to a group.

Treatment Groups:

Group 1: Normal Saline (0.9% Sodium Chloride)

Your child will receive the standard treatment for sepsis, including antibiotics, intravenous fluids, heart function monitoring, mechanical ventilation if needed, and blood pressure medications (vasopressors) if necessary.

Group 2: Ringer's Lactate

In addition to standard sepsis management, your child will receive Ringer's lactate, another commonly used resuscitation fluid in pediatric sepsis.

Group 3: Octaplas LG

In addition to standard sepsis management, your child will receive pharmaceutical synthetic plasma, which contains proteins and essential blood components that have undergone advanced processing to eliminate the risk of infectious disease transmission.

How Many Children Will Participate in This Study? At Fundación Cardioinfantil-Instituto de Cardiología, we are seeking the participation of approximately 150 children in this study.

How Long Will My Child Be in the Study? Your child will remain in their assigned treatment group for up to 28 days from PICU admission or until they no longer require intensive care hospitalization.

DETAILED DESCRIPTION:
Protocol Title: Randomized Clinical Trial Comparing Crystalloids vs. Synthetic Plasma for Fluid Resuscitation in Children with Sepsis - REsuscitation of Sepsis Trial (RESET): Feasibility and Comparative Study

Development Phase: Phase IV Study

Sponsor:

Fundación Cardioinfantil - Instituto de Cardiología Children's Hospital of Pittsburgh - Center for Trauma and Transfusion Medicine Research, University of Pittsburgh, Pittsburgh, USA

Medical Sponsor and International Coordinator Dr. Jaime Fernández - Pediatric Intensivist, Head of the Pediatric Intensive Care Unit, Fundación Cardioinfantil, Bogotá, Colombia Dr. Phillip Spinella, MD, FCCM - Pediatric Intensivist, Department of Surgery and Anesthesia, Children's Hospital of Pittsburgh; Emeritus Professor, Department of Surgery and Critical Care, University of Pittsburgh; Director, Center for Trauma and Transfusion Medicine Research, University of Pittsburgh, Pittsburgh, USA

Drug Manufacturer: Octapharma

Study Center: Fundación Cardioinfantil - Bogotá, Colombia

Study Objectives

Primary Objective:

To evaluate the feasibility in terms of efficacy and safety of crystalloids versus synthetic fresh plasma as the initial resuscitation fluid in children presenting with septic shock. Feasibility study.

Secondary Objectives:

1. Compare hemodynamic parameters using continuous non-invasive cardiac output monitoring (iCON®) between groups.
2. Assess intravascular volume via echocardiography at 6 ± 2, 24 ± 8, and 48 ± 8 hours across groups.
3. Compare the total volume of normal saline, lactate, or plasma administered for resuscitation within the first 6, 24, and 48 hours.
4. Evaluate net fluid balance at 24 and 48 hours.
5. Compare oxygenation parameters (S/F ratio, P/F ratio, oxygenation index) between the two groups at 0, 6, 24, and 48 hours in ventilated children.
6. Assess organ dysfunction scores (PELOD, pSOFA, and NP-MODS) daily for 48 hours.
7. Compare peak inotropic scores daily over 48 hours.
8. Evaluate endothelial injury markers and hemostatic parameters.
9. Assess inflammatory markers and coagulation activation measures.
10. Monitor transfusion-related reactions.
11. Compare healthcare-associated infections.
12. Assess 28-day mortality and cause of death.

Study Design A prospective, randomized, open-label, feasibility-controlled trial.

Investigational Medicinal Product

Patients diagnosed with septic shock who meet the inclusion criteria will be randomly assigned to one of three intervention arms:

* Group A: Bolus dose of 10 mL/kg normal saline (NS) (max. 500 mL) administered over <15 minutes.
* Group B: Bolus dose of 10 mL/kg Ringer's lactate (max. 500 mL) administered over <15 minutes.
* Group C: Pharmaceutical fresh frozen plasma (OCTAPLAS LG®), bolus dose of 10 mL/kg (max. 500 mL) administered over <15 minutes.

The commercial product OCTAPLAS LG® has been registered with INVIMA in Colombia for five years and is used as a plasma replacement in cardiac surgery, hematologic diseases, or intensive care settings where blood bank plasma is unavailable.

Study Population Children aged 1 month to 18 years diagnosed with sepsis, admitted to the Pediatric Intensive Care Unit (PICU) at Fundación Cardioinfantil over a 12-month period, and meeting eligibility criteria.

ELIGIBILITY:
Inclusion criteria

* Age: ≥1 month (corrected gestational age) to 18 years.
* Diagnosis of sepsis with at least one of the following conditions:
* Signs of poor perfusion: prolonged capillary refill ≥2 sec, weak peripheral pulses, unexplained metabolic acidosis (base deficit > (-)5.0 mEq/L), altered. mental status, lactate ≥2 mmol/L (sample drawn without tourniquet use. (Appendix 2). OR
* Systolic blood pressure (SBP) below the 5th percentile for age.
* Signed informed consent from the patient's legal guardian.

Exclusion Criteria:

* Receipt of ≥2 boluses of NS 0.9% or balanced solution in the last 24 hours for the current sepsis episode (bolus defined as ≥10 mL/kg (max. 500 mL) of NS/RL given in <30 min).
* Known allergic reaction to plasma-derived products.
* Known IgA deficiency.
* Suspected or confirmed congestive heart failure.
* Nephrotic syndrome.
* Known chronic kidney disease with fluid overload or congestive heart failure.
* Diagnosed hemorrhagic dengue fever confirmed by antigen or serology (NS1 or IgM positive).

Ages: 4 Weeks to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
Feasibility in terms of efficacy and safety of crystalloids versus synthetic fresh plasma as the initial resuscitation fluid in children presenting with septic shock: Rate of Signed Informed Consent | Within the first 2 hours after presentation to the PICU. Percentage (%)
  Proportion of patients for whom signed informed consent is obtained prior to the intervention.
Feasibility in terms of efficacy and safety of crystalloids versus synthetic fresh plasma as the initial resuscitation fluid in children presenting with septic shock: Time to Plasma Administration | Within the first 24 hours after admission. Minutes (min)
  Time elapsed from clinical indication to administration of the assigned plasma product.
Feasibility in terms of efficacy and safety of crystalloids versus synthetic fresh plasma as the initial resuscitation fluid in children presenting with septic shock: Follow-up Rate | From PICU admission until day 28 or PICU discharge. Percentage (%)
  Proportion of patients with complete follow-up until PICU discharge or day 28, whichever comes first.
Feasibility in terms of efficacy and safety of crystalloids versus synthetic fresh plasma as the initial resuscitation fluid in children presenting with septic shock: Ability to Obtain and Process Biological Samples | During the first 24 hours post-intervention. Percentage (%)
  Percentage of biological samples (for clinical laboratory tests, inflammatory markers, and endothelial biomarkers) successfully collected and processed according to protocol.
Feasibility in terms of efficacy and safety of crystalloids versus synthetic fresh plasma as the initial resuscitation fluid in children presenting with septic shock: Incidence of Clinical Outcomes | Up to 28 days post-intervention or until PICU discharge. Number of events (n), Percentage (%)
  Incidence of clinical outcomes such as mechanical ventilation, inotropic support, multiple organ dysfunction, or mortality.
Efficacy of crystalloids versus synthetic fresh plasma as the initial resuscitation fluid in children presenting with septic shock in clinical variables and supports: Oxygenation as Assessed by PaO₂/FiO₂ Ratio | Within the first 24 hours of intervention. Ratio (unitless)
  Evaluation of oxygenation using the PaO₂/FiO₂ ratio.
Efficacy of crystalloids versus synthetic fresh plasma as the initial resuscitation fluid in children presenting with septic shock in clinical variables and supports: Oxygenation Index (OI) | Within the first 24 hours of intervention. Unitless value
  Oxygenation Index calculated as (FiO₂ × MAP / PaO₂) × 100.
Efficacy of crystalloids versus synthetic fresh plasma as the initial resuscitation fluid in children presenting with septic shock in clinical variables and supports: Intravascular Volume Status | Within the first 24 hours of intervention. Categorized as improved / no change / worsened (qualitative)
  Assessment of intravascular volume status based on clinical and hemodynamic parameters.
Efficacy of crystalloids versus synthetic fresh plasma as the initial resuscitation fluid in children presenting with septic shock in clinical variables and supports: Inotropic Score | Maximum value during the first 24 hours post-intervention. Inotropic score (numeric)
  Quantification of cardiovascular support based on standard inotropic scoring systems.
Efficacy of crystalloids versus synthetic fresh plasma as the initial resuscitation fluid in children presenting with septic shock in clinical variables and supports: Endothelial Injury Markers | Baseline and within 24 hours post-intervention. ng/mL
  Measurement of circulating endothelial biomarkers such as syndecan-1, angiopoietin-2, or others defined in protocol.
Efficacy of crystalloids versus synthetic fresh plasma as the initial resuscitation fluid in children presenting with septic shock in clinical variables and supports: Hemostatic Measures | Baseline and within 24 hours post-intervention. Seconds (for PT/aPTT), mg/dL or ng/mL (as applicable)
  Evaluation of coagulation parameters including PT, aPTT, fibrinogen, and D-dimer levels.
Efficacy of crystalloids versus synthetic fresh plasma as the initial resuscitation fluid in children presenting with septic shock in clinical variables and supports: Incidence of New or Progressive Organ Failure | Up to 28 days post-intervention or until PICU discharge. Number of patients (n), Percentage (%)
  Number of patients with new or worsening organ dysfunction during hospitalization.
Efficacy of crystalloids versus synthetic fresh plasma as the initial resuscitation fluid in children presenting with septic shock in clinical variables and supports: 28-Day All-Cause Mortality | Up to day 28. Number of deaths (n), Percentage (%)
  Death from any cause within 28 days of randomization.
Efficacy of crystalloids versus synthetic fresh plasma as the initial resuscitation fluid in children presenting with septic shock in clinical variables and supports: Cause of Death | Up to 28 days post-randomization. Categorical (by cause)
  Categorization of causes of death (e.g., refractory shock, respiratory failure, neurologic injury).

SECONDARY OUTCOMES:
Compare hemodynamic parameters using continuous non-invasive cardiac output monitoring (iCON®) between groups: Systemic Vascular Resistance (SVR) | During the 24-hour intervention period. dyn·s/cm⁵
  Measurement of systemic vascular resistance using non-invasive cardiac output monitoring (iCON®).
Compare hemodynamic parameters using continuous non-invasive cardiac output monitoring (iCON®) between groups: Cardiac Output (CO) | During the 24-hour intervention period. Liters per minute (L/min)
  Measurement of cardiac output using iCON® monitoring.
Compare hemodynamic parameters using continuous non-invasive cardiac output monitoring (iCON®) between groups: Cardiac Index (CI) | During the 24-hour intervention period. Liters per minute per square meter (L/min/m²)
  Measurement of cardiac index using iCON® monitoring.
Compare hemodynamic parameters using continuous non-invasive cardiac output monitoring (iCON®) between groups: Stroke Volume Variability (SVV) | During the 24-hour intervention period. Percentage (%)
  Measurement of stroke volume variability using iCON® monitoring.
Compare hemodynamic parameters using continuous non-invasive cardiac output monitoring (iCON®) between groups: Pulse Pressure Variation (PPV) | During the 24-hour intervention period. Percentage (%)
  Measurement of pulse pressure variation using iCON® monitoring.
Total Volume of Resuscitation Fluid Administered Within the First 6, 24, and 48 Hours | At 6, 24, and 48 hours after admission. Milliliters (mL)
  Cumulative volume (in milliliters) of the assigned resuscitation fluid (normal saline, lactated Ringer's, or synthetic plasma) administered at three time points: 6 hours, 24 hours, and 48 hours after admission. Volumes will be obtained from the electronic medical records and reported as total volume per patient per time point.
Evaluate endothelial injury markers and hemostatic parameters, and assess inflammatory markers and coagulation activation measures: Plasma Concentration of IL-1 at 0, 6, and 24 Hours | 0, 6, and 24 hours after fluid administration. pg/mL
  Quantification of interleukin-1 (IL-1) in plasma at baseline, 6 hours, and 24 hours post-intervention.
Evaluate endothelial injury markers and hemostatic parameters, and assess inflammatory markers and coagulation activation measures: Plasma Concentration of IL-6 at 0, 6, and 24 Hours | 0, 6, and 24 hours. pg/mL
  Quantification of interleukin-6 (IL-6) in plasma at baseline, 6 hours, and 24 hours.
Evaluate endothelial injury markers and hemostatic parameters, and assess inflammatory markers and coagulation activation measures: Plasma Concentration of IL-10 at 0, 6, and 24 Hours | 0, 6, and 24 hours. pg/mL
  Quantification of interleukin-10 (IL-10) in plasma at baseline, 6 hours, and 24 hours.
Evaluate endothelial injury markers and hemostatic parameters, and assess inflammatory markers and coagulation activation measures: Plasma Concentration of TNF-alpha at 0, 6, and 24 Hours | 0, 6, and 24 hours. pg/mL
  Quantification of tumor necrosis factor alpha in plasma at baseline, 6 hours, and 24 hours.
Evaluate endothelial injury markers and hemostatic parameters, and assess inflammatory markers and coagulation activation measures: Plasma Concentration of Syndecan-1 at 0, 6, and 24 Hours | 0, 6, and 24 hours. ng/mL
  Measurement of endothelial injury marker Syndecan-1.
Evaluate endothelial injury markers and hemostatic parameters, and assess inflammatory markers and coagulation activation measures: Plasma Concentration of Soluble E-selectin (sE-selectin) | 0, 6, and 24 hours. ng/mL
  Measurement of soluble E-selectin levels at 0, 6, and 24 hours.
Evaluate endothelial injury markers and hemostatic parameters, and assess inflammatory markers and coagulation activation measures: Plasma Concentration of Thrombomodulin | 0, 6, and 24 hours. ng/mL
  Measurement of thrombomodulin as a marker of endothelial injury.
Evaluate endothelial injury markers and hemostatic parameters, and assess inflammatory markers and coagulation activation measures: Plasma Concentration of VEGF and VEGFR-1 | 0, 6, and 24 hours. pg/mL
  Quantification of vascular endothelial growth factor (VEGF) and VEGF receptor 1 (VEGFR1) at baseline and post-intervention.
Evaluate endothelial injury markers and hemostatic parameters, and assess inflammatory markers and coagulation activation measures: Plasma Concentration of Coagulation Activation Markers (TAT Complexes, PF-1, PF-2) | 0, 6, and 24 hours. ng/mL
  Measurement of thrombin-antithrombin complexes (TAT), and platelet factor-1 and -2 (PF-1, PF-2) at specified time points.
Safety endpoints, transfusion reactions: Number of Participants with Transfusion-Related Acute Lung Injury (TRALI) | Within 24 hours of intervention. Number of participants
  Incidence of TRALI within 24 hours of resuscitation fluid administration, based on clinical criteria (acute lung injury, hypoxemia, and temporal relationship to transfusion).
Safety endpoints, transfusion reactions: Number of Participants with Transfusion-Associated Circulatory Overload (TACO) | Within 24 hours of intervention. Number of participants
  Incidence of TACO based on clinical signs (e.g., hypertension, pulmonary edema, increased BNP, positive fluid balance) within 24 hours post-transfusion.
Safety endpoints. Transfusion reactions: Number of Participants with Febrile Non-Hemolytic Transfusion Reactions | Within 24 hours of intervention. Number of participants
  Number of febrile non-hemolytic transfusion reactions as defined by unexplained fever during or shortly after transfusion.
Safety endpoints, transfusion reactions: Number of Participants with Allergic Transfusion Reactions | Within 24 hours of intervention. Number of participants
  Incidence of allergic reactions (rash, urticaria, pruritus, or anaphylaxis) occurring within 24 hours of transfusion.

CONTACTS AND LOCATIONS:
Overall Officials: Philp Spinella Dr, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Fundacion CardioInfantil - Instituto de Cardiología, Bogotá, Bogota D.C., Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Iba T, Maier CL, Helms J, Ferrer R, Thachil J, Levy JH. Managing sepsis and septic shock in an endothelial glycocalyx-friendly way: from the viewpoint of surviving sepsis campaign guidelines. Ann Intensive Care. 2024 Apr 24;14(1):64. doi: 10.1186/s13613-024-01301-6. PMID 38658435
- [Background] Obonyo NG, Sela DP, Raman S, Rachakonda R, Schneider B, Hoe LES, Fanning JP, Bassi GL, Maitland K, Suen JY, Fraser JF. Resuscitation-associated endotheliopathy (RAsE): a conceptual framework based on a systematic review and meta-analysis. Syst Rev. 2023 Nov 22;12(1):221. doi: 10.1186/s13643-023-02385-0. PMID 37990333
- [Background] Torres LN, Chung KK, Salgado CL, Dubick MA, Torres Filho IP. Low-volume resuscitation with normal saline is associated with microvascular endothelial dysfunction after hemorrhage in rats, compared to colloids and balanced crystalloids. Crit Care. 2017 Jun 29;21(1):160. doi: 10.1186/s13054-017-1745-7. PMID 28659186